CLINICAL TRIAL: NCT01377740
Title: Non-Invasive Reduction of Abdominal Fat Utilizing the CoolFlex and eZ App 6.3 Applicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA11-001
Record Dates: First submitted 2011-06-16; First posted 2011-06-21 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2012-01

CONDITIONS: Fat Reduction in the Abdomen
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The Zeltiq System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
This study is being performed to reduce unwanted abdominal fat using two different applicators for the Zeltiq System.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the performance of the CoolFlex applicator compared to the performance of the eZ App 6.3 applicator in the treatment of abdominal fat in terms of its ability to achieve a discernable change to the contour of the treated area.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects > 18 years of age and < 65 years of age.
2. Subject has clearly visible fat on the abdomen. (Figure 1)
3. Subject has not had weight change exceeding 10 pounds in the preceding month.
4. Subject agrees to maintain their weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
5. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Subject has had a surgical procedure(s) in the area of intended treatment.
2. Subject has had an invasive fat reduction procedure (e.g., liposuction, abdominoplasty, mesotherapy) in the area of intended treatment.
3. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 6 months.
4. Subject has discernable asymmetry or contour irregularity in the intended treatment area.
5. Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
6. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
7. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
8. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
9. Subject body mass index (BMI) exceeds 40. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
10. Subject is taking or has taken diet pills or supplements within the past month.
11. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation.
12. Subject is pregnant or intending to become pregnant in the next 6 months.
13. Subject is lactating or has been lactating in the past 6 months.
14. Subject is unable or unwilling to comply with the study requirements.
15. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
16. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Independent imaging review | 16 weeks
  The primary effectiveness endpoint is the percent of reviews by the reviewers which either identify no clinically significant difference in fat reduction between the two sides of the abdomen, or identify greater fat reduction on the side of the abdomen treated with the CoolFlex applicator at 8 weeks post-treatment. It is expected that the percentage of reviews identifying no clinically significant difference between the two sides of the abdomen or identifying greater fat reduction on the side of the abdomen treated with the CoolFlex applicator at 8 weeks post-treatment will be at least 75%.

SECONDARY OUTCOMES:
Overall reduction | 16 weeks
  Overall reduction in the fat layer thickness on each side of the abdomen, as demonstrated by comparison of pre-treatment and 8- and 16-week post-treatment ultrasound measurements, for all evaluable subjects (i.e., adequate ultrasound imaging data sets).
Subject satisfaction | 16 weeks
  Subject satisfaction with the Zeltiq procedure as determined by the results of a subject satisfaction questionnaire at the 8- and 16-week follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Boey, MD, Principal Investigator — Arbutus Laser Centre
Locations (2):
- Canada (2):
  - Arbutus Laser Centre, Vancouver, British Columbia
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario

IPD SHARING:
Plan to Share IPD: No